CLINICAL TRIAL: NCT02546999
Title: Does Botulinum Toxin A Make Walking Easier in Children With Cerebral Palsy?
Acronym: WE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); The Hospital of Vestfold (Other); University Hospital of North Norway (Other); Oslo University Hospital (Other); Haukeland University Hospital (Other); Fondation Lenval (Other); Mazowieckie Centrum Neuropsychiatrii, Warszawa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/1195; 2014-002539-32 (EudraCT Number)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy; Muscle Spasticity
Keywords: Botulinum Toxins, Type A; Walking
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- botox (Experimental): Botox® (onabotulinumtoxin A),injections in the calf muscles. The total maximum body dose of Botox® in this study will be 420 Units. Maximum dose per injection site will be 50 Units. The gastrocnemius muscle will receive 5-6 Units Botox® per kg, but maximum 180 Units in each leg. The soleus muscle will receive 2 Units Botox® per kg with maximum dose 60 Units in each leg. Dilution: 100 Units Botox® in 1 ml 0.9% sodium chloride, and the maximum volume per injection site will be 0,5 ml in both study groups. The route of administration is intramuscular injection.
  Interventions: Drug: botox
- placebo (Placebo Comparator): Sterile 0,9% Sodium Chloride injection The placebo dose will be the same dose in ml as the reconstituted Botox
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: botox — The agent will be given only once at point zero in the time scheme for the project.
  Other Names: botulinum toxin A
  Arms: botox
Drug: placebo — The agent will be given only once at point zero in the time scheme for the project.
  Other Names: sodium chloride
  Arms: placebo

SUMMARY:
In Norway, about 60% of all children with cerebral palsy (CP) are being treated with botulinum toxin A (BoNT-A) at 6 years of age, mainly in the legs. Despite this widespread use of the drug, the evidence for a positive effect on walking is insufficient. Moreover, large variation in effect is seen by clinicians. The main objective of the present study is to investigate whether injections with BoNT-A in the calf muscles make walking easier in children with spastic CP within 6 months, reflected by reduced energy cost during walking.

DETAILED DESCRIPTION:
This is an industry independent multicentre clinical trial. The randomization will be done by a computer number random generator and will be carried out and held by the unit of Applied Clinical Research at NTNU. Two strata: age and center.

The study will be conducted according to Consort guidelines and guidelines for Good Clinical Practice. It is approved by the local Ethical committee (REK Nord) and the Norwegian Drug Agency.

Primary research question is: Do BoNT-A injections in the calf muscles make walking easier in children with CP? Secondary research questions: 1) Do BoNT-A injections in the calf muscles increase activity? 2) Do BoNT-A injections in the calf muscles improve walking capacity 3) Do BoNT-A injections in the calf muscles improve perceived performance and satisfaction related to mobility tasks and 4) Do BoNT-A injections in the calf muscles reduce recurrent musculoskeletal pain? The participants will receive the treatment with both local anaesthesia and conscious sedation with oral or nasal benzodiazepines.Outcome measures are made at baseline and 4, 12 and 24 weeks after treatment, with primary endpoint at 12 weeks.

Data will be analyzed using a linear mixed model (LMM). The difference in change in the primary outcome measure (energy cost during walking) between the treated and placebo groups will be done using a post hoc test following the LMM. Secondary, the same model will be used to test for an effect also at 4 and 24 weeks post injection. Age, GMFCS Level, number of prior BoNT-A treatments and study center will be considered as potential covariates.

A substudy will be conducted within the frames of this RCT, aiming to identify characteristics of those who respond to the treatment compared to those who do not respond (outcome measures 6, 7,8 and 9).

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with unilateral or bilateral CP
* GMFCS level I and II
* Signed informed consent
* expected cooperation of the patients for the treatment and follow up.

Exclusion Criteria:

* BoNT-A injections in the lower legs in the last 6 months before intervention
* history of adverse reactions to BoNT-A
* Known hypersensitivity to BoNT-A or to any of the excipients
* Orthopedic surgery in the legs in the last 2 years
* Major cognitive impairments (must be able to take verbal instructions and conduct the test procedure)
* infection at the proposed injection site(s)
* Subclinical or clinical evidence of defective neuromuscular transmission e.g. myasthenia gravis or Lambert-Eaton Syndrome in patients with peripheral motor neuropathic diseases (e.g. amyotrophic lateral sclerosis or motor neuropathy)
* other underlying neurological disorders that may be affected by BoNT-A injections
* Use of aminoglycoside antibiotics or spectinomycin, or other medicinal products that interfere with neuromuscular transmission (e.g. neuromuscular blocking agents)
* Pregnant or breast-feeding
* Childbearing potential not using contraception
* any reason why, in the opinion of the investigator, the patient should not participate
* Children needing deep sedation under treatment

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2015-09; Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Energy cost during walking | 6 months
  Will be measured by a 5 minutes walk test (overground walking at comfortable speed) with simultaneous gas exchange.

SECONDARY OUTCOMES:
Activity | 6 months
  Daily activity, measured by a body worn accelerometer over 4 periods of 7 consecutive days.
Perceived improved performance and satisfaction | 6 months
  Assessed by The Canadian Occupational Performance Measure
Recurrent musculoskeletal pain | 6 months
  Assessed by the Child Health Questionnaire (Norwegian version), and elements from the Brief Pain Inventory (Norwegian version)
Walking capacity | 6 months
  Assessed with OMNI-RPE (OMNI Rating of Perceived Exertion) and a 1 Minute walk test at maximal gait speed

OTHER OUTCOMES:
Gait pattern | 6 months
  3D gait analysis will be carried out on a subset of participants.
Ankle strength | 6 months
  Isometric strength of ankle plantar- and dorsiflexors, will be made on a subset of the participants.
Spasticity | 6 months
  Will be assessed by the use of Tardieu scale. On a subset of participants, concurrent velocity, position and muscle activation will be measured.
Self-perceived effect on walking | 4 weeks
  A qualitative interview will be conducted on a subset of the participants at baseline and post 1 (4 weeks post injection)

CONTACTS AND LOCATIONS:
Overall Officials: Petter Aadahl, md prof, Study Director — St. Olavs Hospital
Locations (7):
- Lenval Foundation Children's Hospital, Nice, France
- Norway (5):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - University Hospital of North-Norway, Tromsø
  - Department of Orthopaedic Surgery, St. Olavs University Hospital, Trondheim
  - Vestfold Hospital trust, Tønsberg
- Mazowieckie Centrum Neuropsychiatrii, Zagorze, Warsaw, Poland

REFERENCES:
- [Background] Braendvik SM, Roeleveld K, Andersen GL, Raftemo AE, Ramstad K, Majkic-Tajsic J, Lamvik T, Lund B, Follestad T, Vik T. The WE-Study: does botulinum toxin A make walking easier in children with cerebral palsy?: Study protocol for a randomized controlled trial. Trials. 2017 Feb 6;18(1):58. doi: 10.1186/s13063-016-1772-8. PMID 28166806
- [Derived] Braendvik SM, Ross Raftemo AE, Roeleveld K, Andersen GL, Ramstad K, Follestad T, Aarli A, Bonikowski M, Vik T; Walking Easier. Does botulinum neurotoxin A make walking easier in children with cerebral palsy? A randomized clinical trial. Dev Med Child Neurol. 2025 Feb;67(2):263-271. doi: 10.1111/dmcn.16038. Epub 2024 Jul 26. PMID 39058740